CLINICAL TRIAL: NCT02535416
Title: A Phase 1, Open-Label Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ARC-520 at Varying Infusion Rates in Normal Adult Volunteers
Brief Title: A Study of ARC-520 at Varying Infusion Rates in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Heparc-1002
Record Dates: First submitted 2015-08-24; First posted 2015-08-28 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — ARC-520; Cetirizine; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- ARC-520 Cohort 1 (Experimental): Single dose, intravenous administration of ARC-520 at 4.0 mg/kg 0.6 mL/min + cetirizine
  Interventions: Drug: ARC-520; Drug: cetirizine
- ARC-520 Cohort 2A (Experimental): Single dose, intravenous administration of ARC-520 at 4.0 mg/kg 0.9 mL/min + cetirizine
  Interventions: Drug: ARC-520; Drug: cetirizine
- ARC-520 Cohort 2 (Experimental): Single dose, intravenous administration of ARC-520 at 4.0 mg/kg 0.75 mL/min + diphenhydramine
  Interventions: Drug: ARC-520; Drug: diphenhydramine
- ARC-520 Cohort 3 (Experimental): Single dose, intravenous administration of ARC-520 at 4.0 mg/kg 0.9 mL/min + diphenhydramine
  Interventions: Drug: ARC-520; Drug: diphenhydramine
- ARC-520 Cohort 4 (Experimental): Single dose, intravenous administration of ARC-520 at 4.0 mg/kg 1.2 mL/min + diphenhydramine
  Interventions: Drug: ARC-520; Drug: diphenhydramine
- ARC-520 Cohort 5 (Experimental): Single dose, intravenous administration of ARC-520 at 4.0 mg/kg 1.5 mL/min + diphenhydramine
  Interventions: Drug: ARC-520; Drug: diphenhydramine
- ARC-520 Cohort 6 (Experimental): Single dose, intravenous administration of ARC-520 at 4.0 mg/kg 5 minute slow bolus push + diphenhydramine
  Interventions: Drug: ARC-520; Drug: diphenhydramine
- ARC-520 Cohort 7 (Experimental): Single dose, intravenous administration of ARC-520 at 5.0 mg/kg 0.9 mL/min + diphenhydramine
  Interventions: Drug: ARC-520; Drug: diphenhydramine
- ARC-520 Cohort 8 (Experimental): Single dose, intravenous administration of ARC-520 at 6.0 mg/kg 0.9 mL/min + diphenhydramine
  Interventions: Drug: ARC-520; Drug: diphenhydramine

INTERVENTIONS:
Drug: ARC-520
Drug: cetirizine
  Arms: ARC-520 Cohort 1; ARC-520 Cohort 2A
Drug: diphenhydramine
  Arms: ARC-520 Cohort 2; ARC-520 Cohort 3; ARC-520 Cohort 4; ARC-520 Cohort 5; ARC-520 Cohort 6; ARC-520 Cohort 7; ARC-520 Cohort 8

SUMMARY:
Single doses of ARC-520 will be evaluated at varying infusion rates and by slow bolus push.

DETAILED DESCRIPTION:
This is a single-center, open-label, sequential cohort, single-dose study of ARC-520 administered intravenously to healthy adult volunteers. Eligible subjects will receive a single intravenous injection of ARC-520. Up to 8 cohorts (a total of approximately 40 subjects) may be enrolled. ARC-520 (4.0 mg/kg) will be administered at increasing infusion rates up to a bolus push in cohort 5. In addition dose levels at 5.0 mg/kg and 6.0 mg/kg will be evaluated at an infusion rate of 0.9 mL/min. For each subject the duration of the study clinic visits is approximately 6 weeks; maximum study duration is approximately 17 weeks including follow-up telephone calls at Days 30, 60 and 90.

Participants will undergo the following evaluations at regular intervals: medical history, physical examinations, bee venom allergy blood test, vital signs measurements, weight, adverse event monitoring, electrocardiograms (ECGs), telemetry, pregnancy test (females), concurrent medication, blood sample collection for hematology, coagulation, chemistry, pharmacokinetics, pharmacodynamics, and drug screens, and urinalysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-55 years of age, inclusive
* Able to provide written informed consent
* BMI between 19.0 and 35.0 kg/m2, inclusive
* 12-lead ECG at Screening and pre-dose with no clinically significant abnormalities
* Highly effective, double barrier contraception (both male and female partners) during the study and for 3 months following the dose of ARC-520
* Willing and able to comply with all study assessments
* Suitable venous access for blood sampling
* Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) and creatinine levels in the normal range
* No abnormal finding of clinical relevance

Exclusion Criteria:

* Pregnant/lactating
* Acute signs of hepatitis/other infection within 4 weeks of Screening
* Concurrent use of anticoagulants, corticosteroids, immunomodulators, or immunosuppressants.
* Use of prescription medication within 14 days prior to study treatment
* Depot injection/implant other than birth control within 3 months of study treatment
* Known diagnosis of diabetes mellitus
* History of autoimmune disease especially autoimmune hepatitis.
* Human immunodeficiency virus (HIV) infection
* Sero-positive for hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Uncontrolled hypertension: blood pressure (BP) > 150/100 mmHg
* History of cardiac rhythm disturbances
* Family history of congenital long QT syndrome, Brugada syndrome or unexplained sudden cardiac death.
* Currently uses medications known to prolong the corrected QT interval (QTc).
* Symptomatic heart failure (per New York Heart Association guidelines)
* Unstable angina, myocardial infarction, severe cardiovascular disease, transient ischemic attack (TIA) or cerebrovascular accident (CVA) within past 6 months
* History of malignancy within last 5 years except for adequately treated basal cell carcinoma, squamous cell skin cancer, superficial bladder tumors, or in situ cervical cancer
* Major surgery within 3 months of Screening
* History of alcohol and/or drug abuse < 12 months from Screening
* Regular use of alcohol within 6 months of Screening
* Evidence of systemic acute inflammation, sepsis or hemolysis.
* Clinically significant psychiatric disorder
* Use of recreational drugs within 3 months of Screening or drugs, such as cocaine, phencyclidine (PCP), and methamphetamines, within 1 year of Screening
* Positive urine drug screen
* History of allergy or hypersensitivity reaction to bee venom
* Positive reaction to the bee venom immunoglobulin E [IgE] test
* Use of investigational agents or devices within 30 days of study dosing or current participation in an investigational study.
* Clinically significant history/presence of any gastrointestinal pathology, unresolved gastrointestinal symptoms, liver or kidney disease
* Cholangitis, cholecystitis, cholestasis, or duct obstruction
* Clinically significant history/presence of neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic, psychiatric, metabolic or other uncontrolled systemic disease
* Blood donation or blood loss (500 mL) within 30 days prior to study treatment
* History of fever within 2 weeks of Screening.
* Excessive exercise/physical activity within 7 days of Screening or enrollment or planned during the study.
* History of coagulopathy, stroke within six (6) months of baseline, and/or concurrent anticoagulant medication(s)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site 1, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2A | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | ARC-520 Cohort 8
Started | 4 | 2 | 4 | 4 | 4 | 4 | 6 | 6 | 6
Completed | 3 | 2 | 4 | 4 | 4 | 4 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Family bereavement overseas | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2A | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | ARC-520 Cohort 8 | Total
Number analyzed (Participants) | 4 | 2 | 4 | 4 | 4 | 4 | 6 | 6 | 6 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.10 (1.49) | 25.96 (7.83) | 29.02 (13.89) | 27.36 (4.91) | 30.05 (9.78) | 28.73 (11.15) | 28.03 (7.79) | 31.19 (11.06) | 31.87 (8.86) | 28.75 (8.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 3 | 3 | 2 | 2 | 5 | 1 | 21
  Male | 2 | 0 | 3 | 1 | 1 | 2 | 4 | 1 | 5 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 1 | 4 | 3 | 4 | 3 | 4 | 5 | 4 | 31
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence that does not necessarily have a causal relationship with this treatment. TEAEs were defined as all AEs starting or worsening after commencement of treatment with investigational product.
Time Frame: post-dose through the end of study (Day 15 ± 1 day) plus 30 days
Population: Safety Population: all enrolled participants
Measure: Number; unit: participants
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2A | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | ARC-520 Cohort 8
Number analyzed (Participants) | 4 | 2 | 4 | 4 | 4 | 4 | 6 | 6 | 6
participants | 2 | 2 | 1 | 3 | 3 | 2 | 5 | 3 | 2

2. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration Versus Time Curve From Zero to 24 Hours (AUC0-24) of the Analytes of ARC-520
Description: Analytes include AD0009 and AD0010 (cholesterol-conjugated siRNA targeting hepatitis B virus [HBV]) and melittin-like peptide (MLP).
Time Frame: Day 1 pre-dose through 48 hours post-dose
Population: All participants with highest achievable infusion rate up to a slow bolus push (Cohort 6) and all participants receiving 4.0, 5.0 and 6.0 mg/kg using an infusion rate of 0.9 mL/min (Cohorts 3, 7 and 8) who had at least one pharmacokinetic (PK) sample collected
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | ARC-520 Cohort 3 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | ARC-520 Cohort 8
Number analyzed (Participants) | 4 | 5 | 6 | 6
ng.hr/mL
  Analyte AD0009 | 350027 (120570) | 331953 (58196) | 403247 (72519) | 605608 (98952)
  Analyte AD0010 | 411580 (131789) | 393161 (64540) | 431980 (69927) | 630774 (87136)
  Analyte MLP | 839718 (181756) | 832929 (132093) | 1015503 (150276) | 1364108 (137352)

3. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration-Time Curve From Time 0 to the Last Quantifiable Plasma Concentration (AUClast) of the Analytes of ARC-520
Description: Analytes include AD0009 and AD0010 (cholesterol-conjugated siRNA targeting HBV) and MLP.
Time Frame: Day 1 pre-dose through 48 hours post-dose
Population: All participants with highest achievable infusion rate up to a slow bolus push (Cohort 6) and all participants receiving 4.0, 5.0 and 6.0 mg/kg using an infusion rate of 0.9 mL/min (Cohorts 3, 7 and 8) who had at least one PK sample collected
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | ARC-520 Cohort 3 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | ARC-520 Cohort 8
Number analyzed (Participants) | 4 | 5 | 6 | 6
ng.hr/mL
  Analyte AD0009 | 361611 (124315) | 340430 (61108) | 416905 (79670) | 638203 (115032)
  Analyte AD0010 | 433632 (139292) | 422964 (72513) | 461601 (84332) | 698567 (107649)
  Analyte MLP | 1022752 (178706) | 1021005 (191504) | 1270330 (195274) | 1722485 (212539)

4. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration Versus Time Curve From Zero Extrapolated to Infinity (AUCinf) of the Analytes of ARC-520
Description: Analytes include AD0009 and AD0010 (cholesterol-conjugated siRNA targeting HBV) and MLP.
Time Frame: Day 1 pre-dose through 48 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | ARC-520 Cohort 3 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | ARC-520 Cohort 8
Number analyzed (Participants) | 4 | 5 | 6 | 6
ng.hr/mL
  Analyte AD0009 | 361820 (124381) | 340591 (61237) | 417153 (79832) | 638965 (115557)
  Analyte AD0010 | 434351 (139573) | 425598 (77283) | 462837 (85266) | 703886 (111074)
  Analyte MLP | 1068557 (160050) | 1080995 (218046) | 1368448 (207758) | 1869597 (282272)

5. Secondary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) of the Analytes of ARC-520
Description: Analytes include AD0009 and AD0010 (cholesterol-conjugated siRNA targeting HBV) and MLP.
Time Frame: Day 1 pre-dose through 48 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ARC-520 Cohort 3 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | ARC-520 Cohort 8
Number analyzed (Participants) | 4 | 5 | 6 | 6
ng/mL
  Analyte AD0009 | 54150 (15711) | 48880 (6155) | 56350 (7516) | 73017 (8532)
  Analyte AD0010 | 49650 (14058) | 46220 (5497) | 49233 (7088) | 64033 (8944)
  Analyte MLP | 76600 (19616) | 75500 (6631) | 85467 (9382) | 112050 (13863)

6. Secondary Outcome: Pharmacokinetics: Clearance (CL) of the Analytes of ARC-520
Description: Analytes include AD0009 and AD0010 (cholesterol-conjugated siRNA targeting HBV) and MLP.
Time Frame: Day 1 pre-dose through 48 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | ARC-520 Cohort 3 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | ARC-520 Cohort 8
Number analyzed (Participants) | 4 | 5 | 6 | 6
mL/hr/kg
  Analyte AD0009 | 12.01 (3.77) | 12.04 (2.05) | 12.40 (2.64) | 9.68 (1.93)
  Analyte AD0010 | 9.92 (3.00) | 9.61 (1.44) | 11.13 (2.17) | 8.72 (1.50)
  Analyte MLP | 3.80 (0.51) | 3.85 (0.91) | 3.73 (0.58) | 3.27 (0.47)

7. Secondary Outcome: Pharmacokinetics: Apparent Volume of Distribution (V) of the Analytes of ARC-520
Description: Analytes include AD0009 and AD0010 (cholesterol-conjugated siRNA targeting HBV) and MLP.
Time Frame: Day 1 pre-dose through 48 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | ARC-520 Cohort 3 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | ARC-520 Cohort 8
Number analyzed (Participants) | 4 | 5 | 6 | 6
mL/kg
  Analyte AD0009 | 70.02 (19.42) | 69.31 (8.53) | 71.49 (9.40) | 62.74 (9.28)
  Analyte AD0010 | 65.98 (18.44) | 71.62 (4.74) | 79.68 (8.52) | 76.21 (12.89)
  Analyte MLP | 58.03 (17.64) | 55.77 (7.25) | 63.92 (9.85) | 56.49 (8.36)

8. Secondary Outcome: Pharmacokinetics: Terminal Elimination Rate Constant (Lambda z) of the Analytes of ARC-520
Description: Analytes include AD0009 and AD0010 (cholesterol-conjugated siRNA targeting HBV) and MLP.
Time Frame: Day 1 pre-dose through 48 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | ARC-520 Cohort 3 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | ARC-520 Cohort 8
Number analyzed (Participants) | 4 | 5 | 6 | 6
1/hr
  Analyte AD0009 | 0.170 (0.027) | 0.170 (0.012) | 0.172 (0.019) | 0.155 (0.021)
  Analyte AD0010 | 0.150 (0.027) | 0.134 (0.025) | 0.140 (0.022) | 0.117 (0.023)
  Analyte MLP | 0.068 (0.015) | 0.070 (0.022) | 0.057 (0.008) | 0.058 (0.013)

9. Secondary Outcome: Pharmacokinetics: Half-Life (t1/2) of the Analytes of ARC-520
Description: Analytes include AD0009 and AD0010 (cholesterol-conjugated siRNA targeting HBV) and MLP.
Time Frame: Day 1 pre-dose through 48 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | ARC-520 Cohort 3 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | ARC-520 Cohort 8
Number analyzed (Participants) | 4 | 5 | 6 | 6
hour
  Analyte AD0009 | 4.10 (0.73) | 4.02 (0.30) | 4.06 (0.44) | 4.56 (0.69)
  Analyte AD0010 | 4.68 (1.03) | 5.31 (1.23) | 5.07 (0.85) | 6.17 (1.34)
  Analyte MLP | 10.41 (2.01) | 10.44 (2.29) | 11.94 (1.32) | 12.24 (2.77)

ADVERSE EVENTS:
Time Frame: post-dose through the end of study (Day 15 ± 1 day) plus 30 days
Description: TEAEs are presented, defined as all AEs starting or worsening after commencement of treatment with investigational product.
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2A | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | ARC-520 Cohort 8
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2 | 0/4 | 0/4 | 0/4 | 0/4 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 0/4 | 0/4 | 0/4 | 0/4 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/4 | 2/2 | 1/4 | 3/4 | 3/4 | 2/4 | 5/6 | 3/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARC-520 Cohort 1 (N=4) | ARC-520 Cohort 2A (N=2) | ARC-520 Cohort 2 (N=4) | ARC-520 Cohort 3 (N=4) | ARC-520 Cohort 4 (N=4) | ARC-520 Cohort 5 (N=4) | ARC-520 Cohort 6 (N=6) | ARC-520 Cohort 7 (N=6) | ARC-520 Cohort 8 (N=6)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdomial discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General symptom (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pustule (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotrasferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No